CLINICAL TRIAL: NCT06129240
Title: An Open-Label ProSpective MultiCENTer Study to Evaluate Safety and Tolerability of Dry Powder Inhaled Treprostinil in Pulmonary Hypertension
Brief Title: An Open-Label ProSpective MultiCENTer Study to Evaluate Safety and Tolerability of Dry Powder Inhaled Treprostinil in PH
Acronym: ASCENT
Status: Active, not recruiting | Type: Observational
Sponsor: Liquidia Technologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LTI-401
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Hypertension; Interstitial Lung Disease
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: PH-ILD
  Interventions: Drug: LIQ861
- Cohort B: PH-ILD
  Interventions: Drug: LIQ861

INTERVENTIONS:
Drug: LIQ861 — trepostinil inhalation powder in combination with inhaler

SUMMARY:
Study LTI-401 is an open-label, multicenter study which will evaluate the safety and tolerability of LIQ861 in subjects who have WHO Group 1 & 3 PH.

DETAILED DESCRIPTION:
Open-label, multicenter study which will evaluate the safety and tolerability of LIQ861 in subjects who have WHO Group 1 & 3 PH.

Cohort A will include approximately 60 subjects who have WHO Group 3 Pulmonary Hypertension associated with interstitial lung disease (PH-ILD)

Cohort B will include approximately 20 subjects who have WHO Group 3 PH-ILD, have been on protocol specified dosing of inhaled treprostinil QID, not at treatment goal, and able to transition to LIQ861.

The primary objective of this study is to evaluate the safety and tolerability of LIQ861 in subjects with WHO Group 1 & 3 Pulmonary Hypertension (PH).

ELIGIBILITY:
Cohort A Key Inclusion Criteria:

1. Males or Females between 18 years to 80 years of age.
2. Has a confirmed diagnosis of WHO Group 3 PH-ILD based on CT chest imaging performed, which demonstrates evidence of diffuse parenchymal lung disease and FEV1/FVC (absolute values) ≥ 70% and are required to have evidence of pulmonary hypertension (PH) as demonstrated from right heart catheterization (RHC) with the following hemodynamic parameters.

   1. i) Pulmonary vascular resistance (PVR) ≥ 3 Wood Units (WU) and ii) Pulmonary capillary wedge pressure (PCWP) of ≤ 15 mmHg and iii) A mean pulmonary arterial pressure (mPAP) of ≥ 30 mmHg.

      OR
   2. An exploratory subset of subjects with ILD: i) Pulmonary vascular resistance (PVR) ≥ 3 Wood Units (WU) and ii) Pulmonary capillary wedge pressure (PCWP) of ≤ 15 mmHg and iii) A mean pulmonary arterial pressure (mPAP) of ≥ 21 mmHg.
3. 6-minute walk distance of ≥ 125 meters

Cohort A Key Exclusion Criteria:

A Subject is not eligible for inclusion in the study if any of the following criteria apply:

1. PH in the Updated WHO Classification Groups 1, 2, 4, or 5.
2. History of hemodynamically significant left-sided heart disease.
3. Exacerbation of underlying lung disease or active pulmonary or upper respiratory infections.
4. Initiation of pulmonary rehabilitation.

Cohort B Key Inclusion Criteria

1. Male or Females between 18 years to 75 years of age at Screening.
2. Has a diagnosis of WHO Group 3 PH-ILD confirmed with CT chest imaging performed at the screening visit, which demonstrates evidence of diffuse parenchymal lung disease and FEV1/FVC (absolute values) ≥70%. Subjects are required to have evidence of pulmonary hypertension (PH) as demonstrated from right heart catheterization (RHC) with the following documented parameters:

   1. Pulmonary vascular resistance (PVR) ≥3 Wood Units (WU) and
   2. Pulmonary capillary wedge pressure (PCWP) of ≤ 15 mmHg and
   3. A mean pulmonary arterial pressure (mPAP) of ≥ 25 mmHg
3. Subjects must be on protocol specified dose of inhaled treprostinil QID not at treatment goal, and able to transition from their prescribed dose of inhaled Treprostinil therapy to LIQ861.
4. 6-minute walk distance of ≥ 200 meters

Cohort B Key Exclusion Criteria

1. PH in the Updated WHO Classification Groups 1, 2, 4, or 5.
2. Inability to titrate inhaled treprostinil above 5 breaths (Tyvaso®) or above 16 mcg Tyvaso DPI®.
3. History of Bronchospasm with Tyvaso or Tyvaso DPI.
4. History of persistent moderate asthma or severe asthma.
5. History of hemodynamically significant left-sided heart disease.
6. Exacerbation of underlying lung disease or active pulmonary or upper respiratory infections.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with PH-ILD
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-02-08 (Estimated)

PRIMARY OUTCOMES:
Cohort A: Incident of treatment-emergent drug/device-related adverse events and Serious Adverse Events (SAEs) | Baseline until the end of the study.
  Treatment-emergent AEs and SAEs will be grouped by MedDRA System Organ Class, dose level at onset, time on drug at onset, and relationship to dose titration. Device-related AEs and SAEs will be grouped by MedDRA System Organ Class, dose level at onset, time on drug at onset, and relationship to dose titration.
Cohort B: Number of participants with treatment-emergent drug/device-related adverse events and Serious Adverse Events (SAEs) | 16 weeks
  Treatment-emergent AEs and SAEs will be grouped by MedDRA System Organ Class, dose level at onset, time on drug at onset, and relationship to dose titration. Device-related AEs and SAEs will be grouped by MedDRA System Organ Class, dose level at onset, time on drug at onset, and relationship to dose titration.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - The Medical Research Group, Inc., Fresno, California
  - UCLA Westwood, Los Angeles, California
  - UC Davis, Sacramento, California
  - UCSF, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Advent Health, Orlando, Florida
  - Tampa General Hospital Center of Research Excellence, Tampa, Florida
  - Vincent Medical Group, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - NYU Langone Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati Health, Cincinnati, Ohio
  - Summit Health, Bend, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist, Houston, Texas
  - University of Utah, Salt Lake City, Utah